CLINICAL TRIAL: NCT02870712
Title: Randomized Controlled Trial of the Effectiveness of Perineal Pain and Security of the Suture Led by the Result of Hemostasis Versus Manual Compression Routine Suture Perineal Tears of First Degree During Childbirth, ImSOLENCE Study
Brief Title: Randomized Controlled Trial of the Effectiveness of Perineal Pain and Security of the Suture Led by the Result of Hemostasis Versus Manual Compression Routine Suture Perineal Tears of First Degree During Childbirth
Acronym: ImSOLENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P/2016/296
Record Dates: First submitted 2016-07-21; First posted 2016-08-17 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2018-09

CONDITIONS: Parturition; Delivery, Obstetric
Keywords: perineal tear of first degree; suture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suture directed (Experimental): The suture of the perineum is headed by obtaining hemostasis by digital compression 5 minutes; If hemostasis is obtained, the perineum will not be sutured. In case of failure of hemostasis, suture of the perineum will be realized.
  Interventions: Procedure: Suture of perineum; Procedure: hemostatis by digital compression
- systematic suture (Active Comparator): systematic suture tears following current recommendations
  Interventions: Procedure: Suture of perineum

INTERVENTIONS:
Procedure: Suture of perineum — suture of the tear to obtain hemostasis
Procedure: hemostatis by digital compression — Digital compression of the tear to obtain hemostasis
  Arms: suture directed

SUMMARY:
During childbirth, the recommendations have evolved to a restriction of episiotomy. This reduction results in an increase of superficial vaginal and perineal tears. These lesions are usually routinely sutured which often causes the onset of discomfort and pain in the immediate postpartum period. Gordon showed, in 1998, improved comfort and pain when the skin was not sutured perineal tears during the second degree. Others have compared different techniques in the same indications (separated points running suture, biological adhesive) without demonstrated impact. These studies were not interested in isolated perineal tears or first degree or the application of a simple manual compression with or without a suture according to the result of hemostasis.

Our objective is to evaluate the possibility of not suture the perineum of the first degree. The use of suture only result of bleeding not yielding to manual compression.

Our approach is guided by the principles of "primum non nocere" and discerning about the dogmatic systematization.

ELIGIBILITY:
Inclusion Criteria:

* single Pregnancy
* primiparae
* delivery by spontaneous vaginal delivery
* forward Delivery (≥ 37 weeks)
* cephalic presentation
* children living
* perineal tear or isolated first-degree vaginal tear

Exclusion Criteria:

* Known haemostatic anomaly
* Premature birth (before 37)
* caesarean
* Instrumental delivery
* Placenta and / or uterine revision
* episiotomy
* perineal tear ≥ 2nd degree

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Composite Outcome Measure for success defined by : - a negligible pain, - satisfactory healing, - no bleeding and infection of the perineum | ten day after childbirth

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided